CLINICAL TRIAL: NCT05564689
Title: Absolute Coronary Flow in Patients With Heart Failure With Reduced Ejection Fraction and Left Bundle Branch Block With Cardiac Resynchronization Therapy
Acronym: FLOW-LBBB
Status: Recruiting | Type: Observational
Sponsor: Ashkan Eftekhari (Other)
Responsible Party: Sponsor-Investigator, Ashkan Eftekhari, Principal Investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: N-20220040
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Left Bundle-Branch Block; Heart Failure; Cardiac Resynchronization Therapy; Dilated Cardiomyopathy
Keywords: absolute coronary flow; fractional flow reserve
MeSH Terms: conditions — Bundle-Branch Block; Heart Failure; Cardiomyopathy, Dilated | interventions — Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with or in need of CRT, left bundle branch block, without ischemic heart disease
  Interventions: Procedure: Intracoronary flow and pressure

INTERVENTIONS:
Procedure: Intracoronary flow and pressure — Measurement of absolute coronary flow and resistance

SUMMARY:
Cardiac resynchronization therapy (CRT) is an effective therapeutic strategy in patients with symptomatic heart failure (HF) patients with LVEF of ≤35% and left bundle branch block (LBBB). However, approximately one-third of CRT-recipients do not improve after therapy (non-responders), despite meeting the required criteria.

Previous studies have documented that the positive respons to CRT is related to the delayed electrical activation of the left ventricle in patients with LBBB. It has also been illustrated that non-ischemic CRT-candidates with LBBB demonstrate lower regional myocardial blood flow and metabolism in the septum. Additionally, it has been suggested that LBBB can lead to impaired coronary blood flow in the left anterior descending artery (LAD). This observation is based on an echocardiography-based study, that showed that the percentage of diastolic flow duration (%DD) in LAD was shorter in patients with LBBB compared to the control-group and patients with right-ventricular pacing.

It has been demonstrated that CRT has positive effects on septal myocardial perfusion in patients with HF and LBBB. The dominant hypothesis explaining this phenomenon is built on improved septal myocardial work after CRT-implantation, which leads to increased myocardial energy and therefore increased myocardial perfusion. In contrast, it has been suggested that due to re-established synchronous left ventricular electrical activation, CRT reduces the septal intramyocardial pressure in early diastole, leading to a relatively longer antegrade flow duration in LAD. Therefore, the aim of the study is to evaluate the effect of CRT on coronary blood flow in LAD in patients with non-ischemic HF and LBBB.

The investigators hypothesize that increased LV-function after CRT not only is due to resynchronized LV ejection and filling, but also improved coronary flow.

The study aims to enroll 60 patients with heart failure due to non-ischemic dilated cardiomyopathy, LBBB, with or without CRT. All patients meeting the criteria will be recruited from the outpatient clinic at the Department of Cardiology, Aalborg University Hospital.

Invasive flow measurements in the LAD, including fractional flow reserve (FFR), absolute coronary flow and -reserve will be conducted with the CRT on and off, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* QRS ≥ 150 ms before implantation
* Heart failure because of dilated cardiomypathy
* Sinus rhythm
* Stable medical therapy
* LBBB
* CRT device

Exclusion Criteria:

* eGFR < 30 ml/min
* Severe valvular heart disease
* Permanent atrial fibrillation or atrial flutter
* Prior PCI or CABG
* Prior myocardial infarction
* Heart failure due to ischemic heart disease
* Other type of device (pacemaker, ICD)
* Not able to give informed consent
* Does not understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with heart failure due to non ischemic dilated cardiomyopathy and LBBB, with or without excisting CRT.
  Eligible patients who are admitted to the Department of Cardiology or at a visit to the outpatient clinic at the Dept. Cardiology Aalborg University Hospital will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Absolute coronary flow | During procedure
  Measurement of absolute coronary flow with/without CRT-function

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Eftekhari, Principal Investigator — Department of Cardiology, Aalborg University Hospital
Locations (1):
- Aalborg Universityhospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided